CLINICAL TRIAL: NCT03430193
Title: Comparative Effectiveness Research of Rehabilitation Methods and Prevention of Refracture After Fractures in Elderly Patients
Brief Title: Fragility Fracture Integrated Rehabilitation Management (FIRM)
Acronym: FIRM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Korea Health Industry Development Institute (Other Government)
Responsible Party: Principal Investigator, Jae-Young Lim, Professor, Department of Rehabilitation Medicine, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HC15C1189
Record Dates: First submitted 2018-01-05; First posted 2018-02-12 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Hip Fractures
Keywords: rehabilitation; multi-disciplinary rehabilitation; clinical pathway; Fragility
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FIRM group (Experimental): FIRM program consisted of total 10 days session including PT, in two times twenty-minute sessions per day and 4 times OT during admission initiated before transfer to rehabilitation ward. PT (Weight bearing exercise, strengthening exercise, gait training, aerobic exercise and functional training) progressed gradually based on individual functional level and OT of activities of daily life (ADL) training (transfer, sit to stand, bed mobility, dressing, self-care retraining and using adaptive equipment) was provided.
  Interventions: Other: FIRM
- Conventional group (Active Comparator): Conventional rehabilitation program consisted of total 10 days session of PT focused on simple standing and gait training, in one time twenty-minute sessions per day.
  Interventions: Other: Conventional rehabilitation
- No-rehabilitation group (No Intervention): Discharged patients not transferred to rehabilitation unit after surgery for hip fracture.

INTERVENTIONS:
Other: FIRM — FIRM program consisted of total 10 days session including PT, in two times twenty-minute sessions per day and 4 times OT during admission initiated before transfer to rehabilitation ward.
  PT (Weight bearing exercise, strengthening exercise, gait training, aerobic exercise and functional training) progressed gradually based on individual functional level and OT of activities of daily life (ADL) training (transfer, sit to stand, bed mobility, dressing, self-care retraining and using adaptive equipment) was provided.
  Arms: FIRM group
Other: Conventional rehabilitation — Conventional rehabilitation program consisted of total 10 days session of PT focused on simple standing and gait training, in one time twenty-minute sessions per day.
  Arms: Conventional group

SUMMARY:
A number of studies for clinical pathway (CP) after hip fracture have been suggested to improve post-fracture outcome. However, CP is not carried out properly in most countries due to inadequate system and awareness, and lack of interdisciplinary approach among orthopaedists, geriatricians and rehabilitation specialists. Thus, we developed Fragility fracture integrated rehabilitation management (FIRM), a new standardized guideline and the multidisciplinary fragility fracture care based on the clinical rehabilitation pathway and conducted a prospective study to evaluate the effects of FIRM compared to conventional rehabilitation.

DETAILED DESCRIPTION:
The purpose of this prospective study

To develop a standardized fragility fracture integrated rehabilitation management (FIRM) based on the critical rehabilitation pathway for fragility fractures.

1. Standardization of initial evaluation for fall and re-fracture risks before rehabilitation
2. Standardization in initial screening for prevention for common complication after fracture and early diagnosis
3. Evidence based standardization in rehabilitation after fragility fracture
4. Development for safe return to normal daily life

ELIGIBILITY:
Inclusion Criteria:

1. Type of fracture : Femoral neck, intertrochanteric, subtrochanteric fracture
2. Type of surgery : Bipolar hemiarthroplasty, THA, ORIF

Exclusion Criteria:

1. Surgery not for hip fracture, but for infection, arthritis, implant loosening, AVN
2. Femur Shaft fracture, acetabular fracture, periprosthetic fracture, pathologic fracture for tumor
3. Combined multiple fracture (ex. Upper extremity)
4. Revision operation
5. Disagree to participation for clinical trial
6. Severe cognitive dysfunction (Obey command ≤1)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2018-02-12 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from baselines mobility status (Functional Ambulatory Category (FAC)) after rehabilitation | 0, 3 month, 6 month, 12 month
  range, 0 to 5; decreasingly worse

SECONDARY OUTCOMES:
Change from baselines mobility status (KOVAL) after rehabilitation | 0, 3 month, 6 month, 12 month
  range, 1 to 7; increasingly worse
Change from baselines mobility status (Functional Independence Measure (FIM)- locomotion) after rehabilitation | 0, 3 month, 6 month, 12 month
  range, 1 to 7; decreasingly worse
Change from baselines balance and fall risk (Berg Balance Scale (BBS)) after rehabilitation | 0, 3 month, 6 month, 12 month
  range, 0 to 56; decreasingly worse
Change from baselines from cognition (Korean Mini-Mental State Examination (K-MMSE)) after rehabilitation | 0, 3 month, 6 month, 12 month
  range, 0 to 30; decreasingly worse
Change from baselines from mood (Korean version of the Geriatric Depression Scale (GDS)) after rehabilitation | 0, 3 month, 6 month, 12 month
  range, 0 to 30 ; increasingly worse
Change from baselines Quality of life (Euro Quality of Life Questionnaire 5-Dimensional Classification (EQ-5D)) after rehabilitation | 0, 3 month, 6 month, 12 month
  range, 0 to 1; decreasingly worse
Change from baselines from activities of daily life (Korean modified Barthel index (K-MBI)) after rehabilitation | 0, 3 month, 6 month, 12 month
  range, 0 to 100; decreasingly worse
Change from baselines from activities of daily life (Korean instrumental ADL (K-IADL)) after rehabilitation | 0, 3 month, 6 month, 12 month
  range, 0 to 3; increasingly worse
Change from baselines frailty (Korean version of fatigue, resistance, ambulation, illnesses, and loss of weight (FRAIL) scale) after rehabilitation | 0, 3 month, 6 month, 12 month
  range, 0 to 5; increasingly worse
Change from baselines hand grip strength after rehabilitation | 0, 3 month, 6 month, 12 month
  measured by a a digital dynamometer (TKK 5401 Grip-D; Takei, Niigata, Japan)

OTHER OUTCOMES:
Mortality | 0, 3 month, 6 month, 12 month
  Mortality rate from number of dead patients among enrolled for the study
Recovery to premorbid ambulatory status | 0, 3 month, 6 month, 12 month
  Comparison premorbid ambulatory status with post-rehabilitation ambulatory status at each follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Young Lim, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beaupre LA, Cinats JG, Senthilselvan A, Lier D, Jones CA, Scharfenberger A, Johnston DW, Saunders LD. Reduced morbidity for elderly patients with a hip fracture after implementation of a perioperative evidence-based clinical pathway. Qual Saf Health Care. 2006 Oct;15(5):375-9. doi: 10.1136/qshc.2005.017095. PMID 17074877
- [Result] Lyons AR. Clinical outcomes and treatment of hip fractures. Am J Med. 1997 Aug 18;103(2A):51S-63S; discussion 63S-64S. doi: 10.1016/s0002-9343(97)90027-9. PMID 9302897
- [Result] Magaziner J, Fredman L, Hawkes W, Hebel JR, Zimmerman S, Orwig DL, Wehren L. Changes in functional status attributable to hip fracture: a comparison of hip fracture patients to community-dwelling aged. Am J Epidemiol. 2003 Jun 1;157(11):1023-31. doi: 10.1093/aje/kwg081. PMID 12777366
- [Result] Sellier E, Labarere J, Sevestre MA, Belmin J, Thiel H, Couturier P, Bosson JL; Association pour la Promotion de l'Angiologie Hospitaliere. Risk factors for deep vein thrombosis in older patients: a multicenter study with systematic compression ultrasonography in postacute care facilities in France. J Am Geriatr Soc. 2008 Feb;56(2):224-30. doi: 10.1111/j.1532-5415.2007.01545.x. Epub 2007 Dec 7. PMID 18070003
- [Result] Hannan EL, Magaziner J, Wang JJ, Eastwood EA, Silberzweig SB, Gilbert M, Morrison RS, McLaughlin MA, Orosz GM, Siu AL. Mortality and locomotion 6 months after hospitalization for hip fracture: risk factors and risk-adjusted hospital outcomes. JAMA. 2001 Jun 6;285(21):2736-42. doi: 10.1001/jama.285.21.2736. PMID 11386929
- [Result] Siu AL, Penrod JD, Boockvar KS, Koval K, Strauss E, Morrison RS. Early ambulation after hip fracture: effects on function and mortality. Arch Intern Med. 2006 Apr 10;166(7):766-71. doi: 10.1001/archinte.166.7.766. PMID 16606814
- [Result] Koval KJ, Cooley MR. Clinical pathway after hip fracture. Disabil Rehabil. 2005 Sep 30-Oct 15;27(18-19):1053-60. doi: 10.1080/09638280500056618. PMID 16278174
- [Result] Halbert J, Crotty M, Whitehead C, Cameron I, Kurrle S, Graham S, Handoll H, Finnegan T, Jones T, Foley A, Shanahan M; Hip Fracture Rehabilitation Trial Collaborative Group. Multi-disciplinary rehabilitation after hip fracture is associated with improved outcome: A systematic review. J Rehabil Med. 2007 Sep;39(7):507-12. doi: 10.2340/16501977-0102. PMID 17724548
- [Result] Adunsky A, Lusky A, Arad M, Heruti RJ. A comparative study of rehabilitation outcomes of elderly hip fracture patients: the advantage of a comprehensive orthogeriatric approach. J Gerontol A Biol Sci Med Sci. 2003 Jun;58(6):542-7. doi: 10.1093/gerona/58.6.m542. PMID 12807926
- [Derived] Lee SY, Beom J, Kim BR, Lim SK, Lim JY; Fragility Fracture Rehabilitation Study Group. Comparative effectiveness of fragility fracture integrated rehabilitation management for elderly individuals after hip fracture surgery: A study protocol for a multicenter randomized controlled trial. Medicine (Baltimore). 2018 May;97(20):e10763. doi: 10.1097/MD.0000000000010763. PMID 29768364